CLINICAL TRIAL: NCT01244386
Title: Low-dose CT Using Iterative Reconstruction in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Responsible Party: Dr Michael M. Maher MD, University College Cork
Other Study IDs: 10-CT-Crohn's
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Computed tomography; Iterative reconstruction; Automatic tube current modulation; Crohn's disease; Inflammatory bowel disease; Radiation dose optimization; C reactive protein
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inflammatory bowel disease: Patients with inflammatory bowel disease requiring CT for clinical purposes will be studied.

SUMMARY:
The purpose of this study is to validate the use of a low-dose computed tomography (CT) protocol and facilitate reduced radiation doses in patients with inflammatory bowel disease (IBD). This is to be achieved using new computer software (Iterative Reconstruction and Automatic Tube Modulation) which will enable low-dose CT imaging at doses equivalent to that of an abdominal radiograph.

DETAILED DESCRIPTION:
The increasing use of CT has prompted the development of new scanning protocols which reduce radiation doses to patients and minimise the likelihood of radiation related morbidity. The use of disease specific low-dose CT examinations is an emerging method of limiting radiation doses.

Research conducted in Cork University Hospital(CUH) by the current authors has identified a pressing need to reduce radiation doses in patients with IBD. A retrospective study of radiation doses in patients with Crohn's disease demonstrated that increasing numbers of CT exams are performed with average cumulative effective doses rising from 7.9 to 25mSv when the first 5-years of the 15 year study period were compared with the final 5-years. Eight-five percent of the dose during the final 5-year period was due to CT. Younger patients with more severe disease requiring surgery or steroids were more likely to undergo an increased number of exams. 15.5% of patients received cumulative effective doses of greater than 75mSv. This quantity of radiation exposure is associated with a 7.3% increase in mortality from cancer. In addition, patients with Crohn's disease are inherently predisposed to gastrointestinal and hepatobiliary carcinoma and small bowel lymphoma.

As an alternative to CT, IBD patients are frequently imaging with conventional abdominal radiography. The effective dose of a conventional abdominal radiograph (CAR) is approximately 10% that of a standard abdominal CT varying between 0.7 -0.1mSv. The current authors have also investigated the value of CAR. We retrospectively examined over 500 CAR's performed over a 16 year period in patients with IBD. Patients had an average of 3.5 CAR's performed but there were positive findings in less than 30% of exams. Many of these findings were non-specific requiring further investigation. For example separation of bowel loops on a plain radiograph has a wide differential diagnosis including abscess formation, presence of a phlegmonous mass, fibrofatty proliferation, bowel wall thickening and lymphadenopathy.

Patients with inflammatory bowel disease referred to CUH will undergo a modified abdominal CT protocol. The radiation dose of a standard CT abdomen and pelvis will be divided into 2 quotients. Patients will have a low-dose CT scan requiring approximately 10% of the dose of a standard abdominal CT. This equates to the radiation dose of a conventional abdominal radiograph. Patients will be imaged with a second CT exam using 90% of the standard abdominal CT dose ensuring a diagnostic study is acquired. Patients will be given oral and intravenous contrast agents as for a standard CT. Patients will have a C-reactive protein measured on the day of CT and will have their heights and weights also measured at the time of scanning. Patients will have a plain film of abdomen performed prior to CT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring a CT abdomen for clinical purposes will be included

Exclusion Criteria:

* Pediatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under the care of the hospital gastrointestinal services including in-patients and outpatients.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The adequacy of low dose CT in patients with Inflammatory bowel disease compared with standard dose CT | At the time of CT
  Radiation dose of a standard CT abdomen and pelvis will be divided into 2 quotients. A low-dose CT scan acquired using automatic tube current modulation (ATM) requiring 10% the dose of a standard abdominal CT and equating to that of a conventional abdominal radiograph. High noise index will be used ensuring reduced mAs. Increased image noise will be overcome by the IR filter. A second CT using 90% of the standard abdominal CT dose will ensure a diagnostic study is acquired.

SECONDARY OUTCOMES:
The correlation of C-reactive protein assay with CT disease severity in inflammatory bowel disease. | CRP sample on same day as CT
  The severity of inflammatory bowel disease will also be quantified based on the CT appearances. The disease severity as measured by CT will be correlated with C-reactive protein measured on the day of imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Maher, MD, Principal Investigator — University College Cork; Owen J O'Connor, MD, Study Director — University College Cork; Fergus Shanahan, MD, Study Director — University College Cork
Locations (1):
- Cork University Hospital, Cork, Co Cork, Ireland

REFERENCES:
- [Background] Desmond AN, O'Regan K, Curran C, McWilliams S, Fitzgerald T, Maher MM, Shanahan F. Crohn's disease: factors associated with exposure to high levels of diagnostic radiation. Gut. 2008 Nov;57(11):1524-9. doi: 10.1136/gut.2008.151415. Epub 2008 Apr 28. PMID 18443021
- [Background] Kalra MK, Rizzo S, Maher MM, Halpern EF, Toth TL, Shepard JA, Aquino SL. Chest CT performed with z-axis modulation: scanning protocol and radiation dose. Radiology. 2005 Oct;237(1):303-8. doi: 10.1148/radiol.2371041227. PMID 16183938
- [Background] Kalra MK, Wittram C, Maher MM, Sharma A, Avinash GB, Karau K, Toth TL, Halpern E, Saini S, Shepard JA. Can noise reduction filters improve low-radiation-dose chest CT images? Pilot study. Radiology. 2003 Jul;228(1):257-64. doi: 10.1148/radiol.2281020606. Epub 2003 May 15. PMID 12750460
- [Background] Kalra MK, Maher MM, Rizzo S, Kanarek D, Shepard JA. Radiation exposure from chest CT: issues and strategies. J Korean Med Sci. 2004 Apr;19(2):159-66. doi: 10.3346/jkms.2004.19.2.159. PMID 15082885
- [Background] O'Connor OJ, Vandeleur M, McGarrigle AM, Moore N, McWilliams SR, McSweeney SE, O'Neill M, Ni Chroinin M, Maher MM. Development of low-dose protocols for thin-section CT assessment of cystic fibrosis in pediatric patients. Radiology. 2010 Dec;257(3):820-9. doi: 10.1148/radiol.10100278. Epub 2010 Sep 27. PMID 20876388